CLINICAL TRIAL: NCT02441933
Title: A Randomized, Multicenter, Open-label, Phase III Trial Comparing Anthracyclines Followed by Taxane Versus Anthracyclines Followed by Taxane Plus Carboplatin as (Neo) Adjuvant Therapy in Patients With Triple-negative Breast Cancer
Brief Title: Carboplatin in EARLY Triple Negative Breast Cancer Trial (PEARLY Trial)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-0074
Record Dates: First submitted 2015-05-04; First posted 2015-05-12 (Estimated); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — taxane; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Active Comparator)
  Interventions: Drug: Taxane
- carboplatin group (Experimental)
  Interventions: Drug: taxane plus carboplatin

INTERVENTIONS:
Drug: taxane plus carboplatin — Doxorubicin (60 mg/m2) IV + cyclophosphamide (600 mg/m2) IV every 3 weeks for 4 cycles followed by taxane plus carboplatin for 4 cycles The taxane plus carboplatin regimen can be selected based on the investigator's discretion from among the following two regimens.
  * Docetaxel (75 mg/m2) IV plus carboplatin (AUC 5) IV every 3 weeks for 4 cycles
  * Paclitaxel (80 mg/m2) IV weekly for 12 doses plus carboplatin (AUC 5) IV every 3 weeks for 4 cycles
  Arms: carboplatin group
Drug: Taxane — Doxorubicin (60 mg/m2) IV + cyclophosphamide (600 mg/m2) IV every 3 weeks for 4 cycles followed by taxane for 4 cycles The taxane regimen can be selected at the investigator's discretion from among the following two regimens.
  * Docetaxel (75 mg/m2) IV every 3 weeks for 4 cycles
  * Paclitaxel (80 mg/m2) IV weekly for 12 doses
  Arms: control group

SUMMARY:
This is a randomized, open-label, multicenter, phase III study comparing anthracyclines followed by taxane to anthracyclines followed by taxane plus carboplatin as (neo)adjuvant therapy in patients with triple-negative breast cancer.

Patients with stage II/III operable triple-negative breast cancer are eligible. Patients who need adjuvant chemotherapy after breast surgery as well as patients who need neoadjuvant chemotherapy for TNBC are eligible.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients who are >18 years of age
2. ECOG 0 or 1
3. The tumor must be invasive carcinoma of the breast on histologic examination
4. The tumor must have been determined to be HER2-negative, as follows:

   * IHC 0 or 1+; or
   * IHC 2+ and ISH non-amplified, with a ratio of <2.0, and if reported, an average HER2 gene copy number of <6 signals/cell; or
   * ISH non-amplified without IHC
5. The tumor must have been determined to be ER- and PR-negative, as assessed by the current ASCO/CAP guidelines.
6. All of the following staging criteria (AJCC 7th edition) must be met:

   * Lymph node-positive disease: cytologically positive in the neoadjuvant group* and pathologically positive in the adjuvant group
   * If the lymph node is cytologically or pathologically negative, the tumor size must be >2.0 cm (* In the neoadjuvant group, if there is evidence of suspicious axillary lymph nodes at the baseline imaging study or physical examination, then FNA or core biopsy is required to confirm the nodal status)
7. The patient must have undergone either a mastectomy or lumpectomy in the adjuvant group
8. The patient must have completed one of the nodal surgery procedures listed below in the adjuvant group:

   * Sentinel lymph node biopsy (SLNB) alone:

V If pathologic nodal staging based on SLNB is pN0 V If pathologic nodal staging based on SLNB is 1 or 2 positive nodes, the primary tumor must be T1 or T2 by pathologic evaluation and lumpectomy and the nodal involvement must be limited to 1 or 2 positive nodes

* SLNB followed by removal of additional non-sentinel LNs if the SLN is positive; or
* Axillary lymphadenectomy with or without SLNB (In the neoadjuvant group, if baseline LN NAB or core biopsy is positive, ALND should be performed) 9) LVEF assessment by echocardiography or MUGA scan must be >50%, regardless of the cardiac imaging facility's lower limit of normal 10) The patient must have adequate hepatic, renal, and bone marrow function;
* Bone marrow function Hb: ≥ 10.0 g/dL ANC: ≥ 1,500/µL Platelet count: ≥ 10 × 10⁴/µL
* Renal function Creatinine: ≤ 1.5 × UNL or Creatine clearance (Ccr) >50 ml/min by the Cockcroft formula
* Hepatic function Total Bilirubin: ≤ 1.5 × UNL AST/ALT: ≤ 2.5 × UNL 10) Ability and willingness to comply with the study visits, treatment, testing, and with the protocol, as per investigator's judgment

Exclusion Criteria:

1. Any prior systemic treatment for primary invasive breast cancer
2. cT4 or pT4 tumors including inflammatory breast cancer
3. Occult breast cancer
4. Evidence of metastatic breast cancer
5. Patients with second primary cancer; EXCEPTIONS: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, DCIS of the breast, thyroid cancer with a size of <2 cm (papillary, follicular, and medullary type), and other solid tumors curatively treated with no evidence of disease for >5 years prior to randomization.
6. Simultaneous bilateral breast cancer
7. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder or uncontrolled infection.
8. Pregnant or breastfeeding women

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 878 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
5-year event-free survival (EFS) | 5 year
  time from Cycle1 Day1 to the occurrence of the following events
  : loco-regional recurrence, distant recurrence, death from any cause, contralateral invasive breast cancer, second primary cancer, and cancer after surgery (not R0 resection), definitive disease progression during neoadjuvant chemotherapy, inoperable status after neoadjuvant chemotherapy

SECONDARY OUTCOMES:
overall survival | 5 year
  Time from C1D1 until death from any cause
Distant recurrence free survival | 5 year
  Time from C1D1 until distant recurrence
loco-regional recurrence free survival | 5 year
  Time from C1D1 until locoregional recurrence
pathologic complete response rate | 5 year
  no evidence of invasive carcinoma in both breast and axillary lymph nodes, regardless of ductal carcinoma in situ (ypT0isN0)

CONTACTS AND LOCATIONS:
Locations (21):
- South Korea (21):
  - Chungbuk university hospital, Cheonju, Chungchung Do
  - National Cancer Center, Goyang, Gyeonggido
  - National Health Insurance Service Ilsan Hospital, Ilsan, Gyeonggido
  - Bundang Cha Hospital, Seongnam, Gyeonggido
  - Ajou universwity Medical Center, Suwon, Gyeonggido
  - Soonchunhyang university Cheonan hospital, Cheonan, Gyungkido
  - Inje University Haeundae Paik Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Seoul national university Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Boramae Medical Center, Seoul
  - Catholic university of Korea, Seoul St. Mary's Hospital, Seoul
  - Chung Ang University Heaelthcare System, Seoul
  - Gangnam Severance hospital, Seoul
  - Korea University Anam hospital, Seoul
  - Kyunghee University Healthcare System, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei Cancer Center at Yonsei University Medical Center, Seoul
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju

REFERENCES:
- [Derived] Kim MH, Kim GM, Ahn JM, Ryu WJ, Kim SG, Kim JH, Kim TY, Han HJ, Kim JY, Park HS, Park S, Park BW, Kim SI, Jeong J, Lee J, Paik S, Kim S, Jung KH, Cho EH, Sohn J. Copy number aberrations in circulating tumor DNA enables prognosis prediction and molecular characterization of breast cancer. J Natl Cancer Inst. 2023 Sep 7;115(9):1036-1049. doi: 10.1093/jnci/djad080. PMID 37166557